CLINICAL TRIAL: NCT02636608
Title: Real World Evidence of the Effectiveness of Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± Ribavirin in Patients With Chronic Hepatitis C - An Observational Study in Hungary - VERITAS
Brief Title: Real World Evidence of the Effectiveness of Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± Ribavirin in Patients With Chronic Hepatitis C - An Observational Study in Hungary
Acronym: VERITAS
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Collaborators: IST GmbH, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-709; HU15-01 (Other: Affiliate Study Tracker Number)
Record Dates: First submitted 2015-12-16; First posted 2015-12-22 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-01

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; Dasabuvir; Paritaprevir/r/Ombitasvir; Observational Study; Quality of Life; Fibrosis; Cirrhosis; Work Ability
MeSH Terms: conditions — Hepatitis C, Chronic; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin: Participants in this observational study received treatment with paritaprevir/ritonavir (r) and ombitasvir with or without dasabuvir ± ribavirin (RBV) for 12 or 24 weeks for the treatment of chronic hepatitis C (CHC), according to hepatitis C virus (HCV) genotype/subtype and stage of liver disease.
  The prescription of treatment regimen was at the discretion of the physician in accordance with local clinical practice and label, was made independently from this observational study and preceded the decision to offer the patient the opportunity to participate in this study.

SUMMARY:
The study seeks to provide evidence of the effectiveness and obtain patient reported outcome (PRO), work productivity and safety data of the interferon-free regimen of paritaprevir (PTV)/ritonavir (r) + ombitasvir (OBV), ± dasabuvir (DSV), ± ribavirin in chronic hepatitis C virus infected participants.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naïve or -experienced adult male or female patients with confirmed chronic hepatitis C (CHC), genotype 1 and 4, receiving combination therapy with the interferon-free paritaprevir (PTV)/ritonavir (r) + ombitasvir (OBV), ± dasabuvir (DSV), ± ribavirin (PTV/r+OBV±DSV±RBV) according to standard of care and in line with the current local label.
* If RBV is co-administered with the PTV/r+OBV±DSV±RBV, it has been prescribed in line with the current local label (with special attention to contraception requirements and contraindication during pregnancy).
* Patients must voluntarily sign and date Subject Information Form and Informed Consent Form prior to inclusion into the study.
* Patient must not be participating or intending to participate in a concurrent interventional therapeutic trial.
* Patient has been started on PTV/r+OBV±DSV±RBV therapy no more than one (1) month prior to the study enrollment.

Exclusion Criteria:

• None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Hepatitis C (CHC)
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2015-11-27 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2018-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ferenci P, Bourgeois S, Buggisch P, Norris S, Curescu M, Larrey D, Marra F, Kleine H, Dorr P, Charafeddine M, Crown E, Bondin M, Back D, Flisiak R. Real-world safety and effectiveness of ombitasvir/paritaprevir/ritonavir +/- dasabuvir +/- ribavirin in hepatitis C virus genotype 1- and 4-infected patients with diverse comorbidities and comedications: A pooled analysis of post-marketing observational studies from 13 countries. J Viral Hepat. 2019 Jun;26(6):685-696. doi: 10.1111/jvh.13080. Epub 2019 Mar 5. PMID 30739368
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This observational study was conducted in 14 medical centers in Hungary experienced in the treatment of chronic hepatitis C (CHC). The first participant entered the study on November 27, 2015 and last patient last visit was on 23 May 2018.
Period: Overall Study
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Started | 244
Received Treatment | 243
Completed (Completed defined as having an HCV RNA assessment performed at least 10 weeks post-treatment) | 233
Not Completed | 11
Not completed — Failure to Return | 4
Not completed — Insufficient Virological Response | 1
Not completed — Death | 3
Not completed — Other | 2
Not completed — Did Not Receive Treatment | 1

BASELINE CHARACTERISTICS:
Population: Treated participants
Groups:
- Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin: Participants in this observational study received treatment with paritaprevir/ritonavir (r) and ombitasvir with or without dasabuvir ± ribavirin (RBV) for 12 or 24 weeks for the treatment of chronic hepatitis C (CHC), according to hepatitis C virus (HCV) genotype/subtype and stage of liver disease.
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 243
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (10.1)
Age, Customized [Count of Participants; unit: Participants]
  18-65 years | 178
  66-84 years | 65
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141
  Male | 102
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 243
Years Since Diagnosis of HCV Infection [Mean (Standard Deviation); unit: years] | 9.2 (7.66)
Hepatitis C Virus Genotype [Count of Participants; unit: Participants]
  Genotype 1a | 9
  Genotype 1a/1b | 5
  Genotype 1b | 227
  Genotype 1b/4 unknown | 1
  Genotype 1 unknown | 1
Cirrhosis Status [Count of Participants; unit: Participants]
  No cirrhosis | 42
  Transition to cirrhosis | 29
  Cirrhosis | 172
Pretreatment Status [Count of Participants; unit: Participants]
  Naive | 83
  Experienced | 160
HCV Ribonucleic Acid (RNA) Level [Mean (Standard Deviation); unit: log10 IU/mL] | 5.79 (0.889)
Assigned Treatment [Count of Participants; unit: Participants] — Treatment regimen was assigned by the physician according to local practice and label. Participants could receive two (paritaprevir/ritonavir and ombitasvir) or three (paritaprevir/ritonavir, ombitasvir, and dasabuvir) direct-acting antiviral (DAA) drugs with or without ribavirin for 12 or 24 weeks.
  Participants
    3 DAA without RBV for 12 weeks | 133
    3 DAA without RBV for 24 weeks | 5
    3 DAA with RBV for 12 weeks | 96
    3 DAA with RBV for 24 weeks | 9
Co-morbidities [Count of Participants; unit: Participants]
  Any co-morbidity or co-infection | 197
  Co-infections | 1
  Hepatitis B | 1
  Liver and/or CHC related co-morbidities | 47

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virological Response 12 Weeks Post-treatment (SVR12)
Description: Sustained virologic response was defined as hepatitis C virus ribonucleic acid (HCV RNA) levels less than 50 IU/mL 12 weeks after the last dose of study drug. Participants with missing HCV RNA were counted as virological failure.
Time Frame: 12 weeks after the last dose of study drug (week 24 or 36 depending on the treatment regimen)
Population: The Core population, defined as enrolled participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 238
percentage of participants | 94.5 [90.9 to 96.8]

2. Secondary Outcome: Percentage of Participants With Sufficient Follow-up Who Achieved Sustained Virological Response 24 Weeks Post-treatment (SVR24)
Description: Sustained virologic response was defined as hepatitis C virus ribonucleic acid (HCV RNA) levels less than 50 IU/mL 24 weeks after the last dose of study drug.
  The Core population with sufficient follow-up data regarding SVR24 included all core population participants who
  * had evaluable HCV RNA data ≥ 126 days after the last actual dose of the ABBVIE REGIMEN
  * or a HCV RNA value ≥ 50 IU/mL at the last measurement post-baseline
  * or had HCV RNA < 50 IU/mL at the last measurement post-baseline, but no HCV RNA measurement ≥ 126 days after the last actual dose of the ABBVIE REGIMEN due to reasons related to safety (e.g. dropped out due to adverse event) or virologic failure.
Time Frame: 24 weeks after the last dose of study drug (week 36 or 48 depending on the treatment regimen)
Population: The Core population with sufficient follow-up data regarding SVR24
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 232
percentage of participants | 96.6 [93.3 to 98.2]

3. Secondary Outcome: Percentage of Participants Achieving Virological Response at End of Treatment
Description: Virologic response was defined as hepatitis C virus ribonucleic acid (HCV RNA) levels less than 50 IU/mL.
Time Frame: End of treatment (week 12 or 24 depending on the treatment regimen)
Population: The Core population defined as enrolled participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 238
percentage of participants | 97.1 [94.1 to 98.6]

4. Secondary Outcome: Percentage of Participants With Relapse
Description: Relapse was defined as participants with a virologic response (VR; HCV RNA < 50 IU/mL) at end of treatment (EOT) followed by HCV RNA ≥ 50 IU/mL at any time after the end of treatment.
Time Frame: End of treatment (week 12 or 24 depending on the treatment regimen) and up to 24 weeks after the end of treatment.
Population: The Core population with VR at EOT, who completed treatment, and had ≥ 1 HCV RNA measurement ≥ 70 days post-treatment or were a treatment failure between EOT and day 70.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 225
percentage of participants | 1.3 [0.5 to 3.8]

5. Secondary Outcome: Number of Participants With Breakthrough
Description: Breakthrough was defined as at least one documented HCV RNA < 50 IU/mL followed by HCV RNA ≥ 50 IU/mL during treatment.
Time Frame: 12 or 24 weeks (depending on the treatment regimen)
Population: The Core population with at least one documented HCV RNA < 50 IU/mL while on treatment and at least one on-treatment or EOT measurement thereafter.
Measure: Count of Participants; unit: Participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 8
Participants | 0

6. Secondary Outcome: Percentage of Participants in Each Non-response Category 12 Weeks Post-treatment
Description: SVR12 non-response was categorized according to the following:
  * On-treatment virologic failure (breakthrough [at least one documented HCV RNA < 50 IU/mL followed by HCV RNA ≥ 50 IU/mL during treatment] or failure to suppress [each measured on-treatment HCV RNA value ≥ 50 IU/mL]);
  * Relapse, defined as HCV RNA < 50 IU/mL at EOT followed by HCV RNA ≥ 50 IU/mL post-treatment in patients who completed treatment (not more than 7 days shortened);
  * Death;
  * Premature treatment discontinuation with no on-treatment virologic failure;
  * None of the above criteria or missing SVR12 data
Time Frame: 12 weeks after the last dose of study drug (week 24 or 36 depending on the treatment regimen)
Population: The Core population
Measure: Count of Participants; unit: Participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 238
Participants
  On-treatment virologic failure | 2
  Relapse | 3
  Death | 3
  Premature treatment discontinuation | 2
  None of the above criteria | 3

7. Secondary Outcome: Percentage of Participants With Adherence to the ABBVIE Regimen, by Adherence Category
Description: Adherence to the ABBVIE treatment regimen is expressed as a percentage of the target dose and was calculated as:
  Cumulative dose taken / (initial prescribed dose * planned duration) * 100
  The ABBVIE regimen consists of paritaprevir/r and ombitasvir with or without dasabuvir.
Time Frame: From first dose of study drug to end of treatment, 12 to 24 weeks depending on the treatment regimen.
Population: Core population
Measure: Number; unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 238
percentage of participants
  > 105% | 3.4
  > 95% to ≤ 105% | 93.7
  > 80% to ≤ 95% | 0.8
  > 50% to ≤ 80% | 0.8
  ≤ 50% | 1.3

8. Secondary Outcome: Percentage of Participants With Adherence to Ribavirin by Adherence Category
Description: Adherence to ribavirin is expressed as a percentage of the target dose, and was calculated as:
  Cumulative dose taken / (initial prescribed dose * planned duration) * 100
Time Frame: From first dose of study drug to end of treatment, 12 to 24 weeks depending on the treatment regimen
Population: Core population who were prescribed ribavirin
Measure: Number; unit: percentage of participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 105
percentage of participants
  > 105% | 1.0
  > 95% to ≤ 105% | 78.1
  > 80% to ≤ 95% | 5.7
  > 50% to ≤ 80% | 6.7
  ≤ 50% | 8.6

9. Secondary Outcome: Percentage of Ribavirin Treatment Days in Relation to the Target Number of Ribavirin Treatment Days
Time Frame: From first dose of study drug to end of treatment, 12 to 24 weeks depending on the treatment regimen.
Population: Core population who were prescribed ribavirin
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 105
percentage of days | 93.1 (22.20)

10. Secondary Outcome: Number of Participants Who Received Concomitant Medications
Description: Concomitant medication other than for chronic hepatitis C used from the time when the decision was made to initiate treatment with paritaprevir/ritonavir and ombitasvir with or without dasabuvir until after the last dose.
Time Frame: From first dose of study drug to end of treatment, 12 to 24 weeks depending on the treatment regimen
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 243
Participants
  Any concomitant medication | 169
  Beta blocking agents | 78
  ACE inhibitors | 53
  Diuretics | 42
  Peptic ulcer / gastro-oesophageal reflux disease | 42
  Calcium channel blockers | 34
  Blood glucose-lowering drugs | 27
  Mineral supplements | 25

11. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events, or Pregnancies
Time Frame: From first dose of study drug through 30 days after last dose (16 or 28 weeks depending on the treatment regimen)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 243
Participants
  Adverse events | 29
  Serious adverse events | 6
  Pregnancies | 0

12. Secondary Outcome: Change From Baseline in EuroQol 5 Dimension 5 Level (EQ-5D-5L) VAS Score
Description: The EQ-5D-5L is a health state utility instrument that evaluates preference for health status. The 5 items in the EQ-5D-5L comprise 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each of which are rated on 5 levels of severity (1: indicating no problem, 2: indicating slight problems, 3: indicating moderate problems, 4: indicating severe problems, 5: indicating extreme problems), and a separate visual analog scale (VAS).
  The VAS assesses overall health on a scale from 0 (worst health imaginable) to 100 (best health imaginable). The higher the score the better the health status.
Time Frame: Baseline, end of treatment (week 12 or 24 depending on the treatment regimen), and at 12 and 24 weeks after end of treatment
Population: Core population with available data at baseline and each time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV: Participants received paritaprevir/ritonavir, ombitasvir, and dasabuvir without ribavirin for 12 or 24 weeks.
- Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir With RBV: Participants received paritaprevir/ritonavir, ombitasvir, and dasabuvir with ribavirin for 12 or 24 weeks.
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir With RBV
Number analyzed (Participants) | 128 | 102
units on a scale
  End of treatment: number analyzed (Participants) | 121 | 97
  End of treatment | 5.70 [3.19 to 8.21] | 2.77 [-0.03 to 5.57]
  12 weeks after end of treatment: number analyzed (Participants) | 113 | 86
  12 weeks after end of treatment | 9.18 [6.83 to 11.5] | 5.98 [3.29 to 8.67]
  24 weeks after end of treatment: number analyzed (Participants) | 119 | 93
  24 weeks after end of treatment | 10.5 [8.04 to 13.0] | 6.07 [3.26 to 8.87]

13. Secondary Outcome: Change From Baseline in EuroQol 5 Dimension 5 Level (EQ-5D-5L) Index Score
Description: The EQ-5D-5L is a health state utility instrument that evaluates preference for health status. The 5 items in the EQ-5D-5L comprise 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each of which are rated on 5 levels of severity (1: indicating no problem, 2: indicating slight problems, 3: indicating moderate problems, 4: indicating severe problems, 5: indicating extreme problems), and a separate visual analog scale (VAS).
  Responses to the 5 dimension scores were combined and converted into a single preference-weighted health utility index score by applying country-specific weights.The range for EQ-5D-5L index score is 0 to 1 where '0' is defined as a health state equivalent to being dead and '1' is full health.The higher the score the better the health status.
Time Frame: as for outcome 12
Population: Core population with available data at baseline and each time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir With RBV
Number analyzed (Participants) | 124 | 103
units on a scale
  End of treatment: number analyzed (Participants) | 115 | 96
  End of treatment | 0.02 [-0.00 to 0.03] | 0.02 [-0.00 to 0.04]
  12 weeks after end of treatment: number analyzed (Participants) | 108 | 85
  12 weeks after end of treatment | 0.03 [0.01 to 0.05] | 0.04 [0.02 to 0.06]
  24 weeks after end of treatment: number analyzed (Participants) | 114 | 94
  24 weeks after end of treatment | 0.04 [0.02 to 0.06] | 0.04 [0.02 to 0.06]

14. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Absenteeism
Description: The WPAI Hepatitis C V2.0 is an HCV specific questionnaire used to measure work absenteeism, work presenteeism, and daily activity impairment. Respondents were asked about time missed from work and time while at work during which productivity was impaired in the past seven days. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity.
  Absenteeism indicates the percentage of work time missed due to health problems.
Time Frame: as for outcome 12
Population: The Core population who were employed and with available data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 68
percent impairment
  End of treatment: number analyzed (Participants) | 64
  End of treatment | -2.1 (21.6)
  12 weeks after end of treatment: number analyzed (Participants) | 59
  12 weeks after end of treatment | -1.7 (22.2)
  24 weeks after end of treatment: number analyzed (Participants) | 66
  24 weeks after end of treatment | 1.0 (19.6)

15. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Presenteeism
Description: The WPAI Hepatitis C V2.0 is an HCV specific questionnaire used to measure work absenteeism, work presenteeism, and daily activity impairment. Respondents were asked about time missed from work and time while at work during which productivity was impaired in the past seven days. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity.
  Presenteeism indicates the percentage of impairment while working due to health problems.
Time Frame: as for outcome 12
Population: The Core population who were employed and with available data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 81
percent impairment
  End of treatment: number analyzed (Participants) | 67
  End of treatment | 0.6 (28.8)
  12 weeks after end of treatment: number analyzed (Participants) | 61
  12 weeks after end of treatment | -5.7 (25.1)
  24 weeks after end of treatment: number analyzed (Participants) | 67
  24 weeks after end of treatment | -7.3 (23.3)

16. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Total Work Productivity Impairment (TWP)
Description: The WPAI Hepatitis C V2.0 is an HCV specific questionnaire used to measure work absenteeism, work presenteeism, and daily activity impairment. Respondents were asked about time missed from work and time while at work during which productivity was impaired in the past seven days. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity.
  Total work productivity impairment (TWP) indicates the percentage of overall work impairment due to health problems.
Time Frame: as for outcome 12
Population: The Core population who were employed and with available data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 78
percent impairment
  End of treatment: number analyzed (Participants) | 62
  End of treatment | -2.3 (34.5)
  12 weeks after end of treatment: number analyzed (Participants) | 58
  12 weeks after end of treatment | -8.1 (30.5)
  24 weeks after end of treatment: number analyzed (Participants) | 65
  24 weeks after end of treatment | -7.3 (27.3)

17. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Total Activity Impairment
Description: The WPAI Hepatitis C V2.0 is an HCV specific questionnaire used to measure work absenteeism, work presenteeism, and daily activity impairment. Respondents were asked about time missed from work and time while at work during which productivity was impaired in the past seven days. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity.
  Total activity impairment (TAI) indicates the percentage of general (non-work) activity impairment due to health problems.
Time Frame: as for outcome 12
Population: The Core population with available data at baseline and each time point.
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 194
percent impairment
  End of treatment: number analyzed (Participants) | 177
  End of treatment | -0.5 (29.4)
  12 weeks after end of treatment: number analyzed (Participants) | 157
  12 weeks after end of treatment | -6.7 (28.4)
  24 weeks after end of treatment: number analyzed (Participants) | 170
  24 weeks after end of treatment | -8.5 (26.6)

18. Secondary Outcome: Change From Baseline in Patient Activation Measure 13 (PAM-13)
Description: PAM-13 is a measure used to assess the patient knowledge, skill, and confidence for self-management, consisting of 13 questions. Each of the 13 items can be answered with one of four possible response options, which are "disagree strongly" (1), "disagree" (2), "agree" (3), "agree strongly" (4). Scores were summed to calculate the overall raw score, then transformed to a scale with a theoretical range 0 to 100, based on calibration tables, with higher PAM scores indicating that the participant is likely to participate more actively in health care processes and takes more responsibility for his or her health.
Time Frame: Baseline and end of treatment (week 12 or 24 depending on the treatment regimen)
Population: The Core population with available data at baseline and end of treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir With RBV
Number analyzed (Participants) | 98 | 90
units on a scale | 0.85 [-1.04 to 2.73] | 0.22 [-1.75 to 2.19]

19. Secondary Outcome: Number of Participants Who Participated in the AbbVie Patient Support Program (PSP)
Time Frame: Up to post treatment week 24
Population: Core population
Measure: Count of Participants; unit: Participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 238
Participants | 179

20. Secondary Outcome: Utilization of the AbbVie Patient Support Program (PSP) Components
Description: At the end of treatment visit participants were asked to indicate which of the following PSP services they had used:
  * Personal support (e.g., Care Coach)
  * Printed educational material
  * Online educational materials
  * Web-portal
  * App
Time Frame: End of treatment (week 12 or 24 depending on the treatment regimen)
Population: Core population who participated in the PSP
Measure: Count of Participants; unit: Participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 179
Participants
  Any | 141
  Personal support | 134
  Printed educational material | 128
  Online educational material | 58
  Web-portal | 65
  App | 54
  None/missing | 38

21. Secondary Outcome: Satisfaction With the AbbVie Patient Support Program (PSP) Components
Description: At the end of treatment visit participants were asked to indicate their level of satisfaction with each of the PSP services they had used.
Time Frame: End of treatment (weeks 12 or 24 depending on treatment regimen)
Population: Core population who participated in the PSP with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 179
Participants
  Personal support: number analyzed (Participants) | 134
  Personal support: Very good | 95
  Personal support: Good | 33
  Personal support: Satisfactory | 6
  Personal support: Poor | 0
  Printed educational material: number analyzed (Participants) | 104
  Printed educational material: Very good | 50
  Printed educational material: Good | 42
  Printed educational material: Satisfactory | 11
  Printed educational material: Poor | 1
  Online educational material: number analyzed (Participants) | 56
  Online educational material: Very good | 21
  Online educational material: Good | 27
  Online educational material: Satisfactory | 8
  Online educational material: Poor | 0
  Web-portal: number analyzed (Participants) | 56
  Web-portal: Very good | 24
  Web-portal: Good | 23
  Web-portal: Satisfactory | 8
  Web-portal: Poor | 1
  App: number analyzed (Participants) | 47
  App: Very good | 14
  App: Good | 31
  App: Satisfactory | 2
  App: Poor | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 30 days after last dose (16 to 28 weeks depending on treatment regimen)
Groups:
- Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV: Participants received paritaprevir/ritonavir, ombitasvir, and dasabuvir without ribavirin for12 or 24 weeks.
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir With RBV
All-Cause Mortality (participants affected / at risk) | 0/138 | 3/105
Serious Adverse Events (participants affected / at risk) | 3/138 | 4/105
Other Adverse Events (participants affected / at risk) | 0/138 | 16/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV (N=138) | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir With RBV (N=105)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
HOSPITALISATION (Surgical and medical procedures) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir Without RBV (N=138) | Paritaprevir/Ritonavir + Ombitasvir + Dasabuvir With RBV (N=105)
ANAEMIA (Blood and lymphatic system disorders) | NA | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2015-08-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT02636608/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT02636608/SAP_001.pdf